CLINICAL TRIAL: NCT02384746
Title: Phase I Study of the Combination of MLN9708 and Fulvestrant in Patients With Advanced Estrogen Receptor Positive Breast Cancer
Brief Title: Phase I Study of the Combination of MLN9708 and Fulvestrant
Acronym: Millennium
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gary Schwartz, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D13036
Record Dates: First submitted 2014-11-20; First posted 2015-03-10 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: metastatic breast cancer; ER-positive; HER2-negative; Fulvestrant; MLN9708
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combination Treatment (Experimental): Fulvestrant (500mg) + MLN9708 (2.3, 3, and 4mg)
  Interventions: Drug: Fulvestrant; Drug: MLN9708

INTERVENTIONS:
Drug: Fulvestrant — 500 mg intramuscular every 28 days
  Other Names: Faslodex
Drug: MLN9708 — Subjects will be treated in 3 dose cohorts of MLN9708, at 2.3, 3, and 4 mg orally on days 1, 4, 8, and 11 every 21 days.
  Other Names: Ixazomib

SUMMARY:
Participants in this study will have been diagnosed with advanced breast cancer that has become worse while being treated with fulvestrant. Participants will have estrogen-receptor positive disease, and have completed menopause.

There is information from research labs which suggests that drugs that work like MLN9708 help kill breast cancer cells that have been treated with fulvestrant. The purpose of the study is to determine the proper dose as well as the good and bad effects of MLN9708 when it is given in combination with fulvestrant. The Investigators also want to learn more about how the drug combination affects tumor cells.

The amount of MLN9708 participants receive will be determined by when they enter this study. Three different doses will be given to different participants. The Investigators expect to enroll a total of 12-18 people.

DETAILED DESCRIPTION:
Subjects with metastatic ER+/HER2- breast cancer with disease progression on Fulvestrant, for whom continuation of endocrine therapy would be an appropriate treatment, will be treated with the combination of MLN9708 (proteasome inhibitor) and Fulvestrant (anti-estrogen). Subjects with visceral or soft tissue disease will have a tumor biopsy while on treatment with Fulvestrant but prior to initiation of MLN9708 to confirm ER/PR/HER2 status, and to provide a baseline specimen for molecular analysis. A biopsy of the same tumor will be obtained after 2 days of treatment with MLN9708 plus Fulvestrant (i.e. on day 3). Patients with bone-only disease will be eligible for the study, but will not be biopsied.

The Investigators propose a 3x3 dose-escalation trial to assess the safety and efficacy of Fulvestrant and three dose levels of MLN9708 (2.3, 3, and 4mg) Subjects will be treated with Fulvestrant (500mg) once every four weeks on day 1. The dose of MLN9708 will start at 2.3mg, which is about 50% of the phase 3 dose in another ongoing study. If 2.3mg MLN9708 does not induce any grade 3 non-hematologic toxicity, or any grade 4 hematologic toxicity by CTCAE v4.0 (Common Terminology Criteria for Adverse Events, version 4.0) in any of the 3 subjects treated for 1 cycle, the Investigators will treat another 3 subjects with the combination of Fulvestrant and MLN9708 (3mg); and if no grade 3 non-hematologic toxicity, or any grade 4 hematologic toxicity by CTCAE v4.0 is seen over the first cycle, the Investigators will treat another 3 subjects with Fulvestrant and MLN9708 (4mg, which is the phase 3 dose). If dose-limiting toxicity is observed in 1/3 subjects, the Investigators will treat an additional 3 subjects at that same dose. If dose-limiting toxicity is seen in 2 of 6 subjects at any dose level, that dose level will be considered the maximum tolerated dose, and a total of 6 subjects will be treated at the prior dose. Plasma pharmacokinetic profiles of MLN9708 will be determined over 21 days after the first dose of the combination.

Pre- and post- treatment tumor biopsies will be formalin-fixed and paraffin-embedded. Tissue sections will be analyzed by H&E (Hematoxylin and eosin) staining and immunohistochemistry using antibodies against markers of proliferation, apoptosis, estrogen receptor alpha activation, endoplasmic reticulum stress, and polyubiquitin. Proteasome activity of whole blood will be determined using samples acquired prior to treatment initiation, and on day 3. Tumor-specific plasma DNA will also be measured prior to treatment initiation and after the first two doses of MLN9708.

ELIGIBILITY:
Inclusion Criteria:

1. Female post-menopausal patients 18 years or older. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
2. Patients must have either A) histologic documentation of metastatic or locally advanced breast cancer by needle or incisional biopsy, or B) history of breast cancer with radiologic evidence of bone-only metastatic disease.
3. Patients must be post-menopausal based on either a history of an oophorectomy, or at lease one year of amenorrhea. An elevated serum gonadotropin level can be used to confirm menopausal status in a subject with one year or more of amenorrhea.
4. The invasive cancer must be HER2-negative, defined as IHC0-1+, or with a FISH ratio of <1.8 if IHC is 2+ or if IHC has not been performed.
5. Metastatic or locally advanced breast cancer for which endocrine therapy is an appropriate treatment option.
6. Patients must have been treated with Fulvestrant for at least 56 days as their most recent anti-cancer treatment, and they must be tolerating Fulvestrant with at most grade I toxicity by CTCAE v4.0.
7. Disease progression based on RECIST criteria while the subject has been taking Fulvestrant, and for which continuation of endocrine therapy would be appropriate.
8. The subject must agree to undergo pre- and post- treatment research biopsies if a non-osseous metastatic site is available for biopsy.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
10. Life expectancy 6 months or longer.
11. Patients must meet the following clinical laboratory data:

    * Absolute Neutrophil Count (ANC) ≥ 1,000/mm(3) and platelet count ≥75,000/mm(3)
    * Total bilirubin ≤ 1.5 x the upper limit of normal range (ULN).
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN.
    * Calculated creatinine clearance ≥ 30 mL/min
12. Ability to give informed consent.

Exclusion Criteria:

1. Failure to have fully recovered (i.e., ≤ Grade 1 toxicity) from the reversible effects of prior chemotherapy or endocrine therapy, except for Grade 2 or greater anemia.
2. Major surgery within 14 days before enrollment.
3. Radiotherapy within 14 days before enrollment. If the involved field is small, 7 days will be considered a sufficient interval between treatment and administration of the MLN9708.
4. Central nervous system involvement.
5. Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
6. Evidence of current uncontrolled cardiovascular conditions.
7. Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2 or CYP3A, or strong inducers of CYP3A.
8. Ongoing or active systemic infection, active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
9. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
10. Known allergy to any of the study medication, their analogues, or excipients in the various formulations of any agent.
11. Known gastrointestinal (GI) disease or GI procedure that could interfere with oral absorption or tolerance of MLN9708 including difficulty swallowing.
12. Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have evidence of residual disease.
13. Patient has ≥ grade 3 peripheral neuropathy, or grade 2 with pain on clinical examination during the screening period.
14. Participation in other clinical trials within 21 days of the start of this trial or throughout the duration of this trial.
15. Visceral crisis or rapidly progressive disease for which chemotherapy would be indicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events prior to commencing a second cycle of treatment. | End of cycle one - Day 21 of Cycle 1
  If the current dose of MLN9708 does not induce any grade 3 non-hematologic toxicity, or any grade 4 hematologic toxicity in any of 3 subjects treated for one cycle, another 3 participants will be treated at the next dose level of MLN9708 (up to 4mg, which is the current phase 3 dose)

SECONDARY OUTCOMES:
Time to Disease Progression | First assessment on Day 1 Cycle 3 - After two cycles, or 42 days of treatment, and then reassessed every 2 cycles or 42 days thereafter
  The length of time on study until there is evidence of disease progression by Response Evaluation Criteria in Solid Tumors (Recist) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Schwartz, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Schwartz G, Shee K, Romo B, Marotti J, Kisselev A, Lewis L, Miller T. Phase Ib Study of the Oral Proteasome Inhibitor Ixazomib (MLN9708) and Fulvestrant in Advanced ER+ Breast Cancer Progressing on Fulvestrant. Oncologist. 2021 Jun;26(6):467-e924. doi: 10.1002/onco.13733. Epub 2021 Mar 18. PMID 33641211